CLINICAL TRIAL: NCT02191007
Title: Multi-center,Single Blind, Parallel-Controlled Study of the Efficacy and Safety of Calcipotriol Betamethasone Ointment Plus Calcipotriol Ointment in Sequential Therapy to Psoriasis Vulgaris
Brief Title: Efficacy and Safety Study of Calcipotriol Betamethasone Plus Calcipotriol in Sequential Therapy to Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, xjpfW, Wang Gang, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CUP2012D001
Record Dates: First submitted 2013-12-26; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Calcipotriol/Betamethasone and Calcipotriol (Experimental): Calcipotriol/Betamethasone ointment 1/d for 4 weeks; Calcipotriol ointment bid for 6 weeks on-demand treatment period;
  Interventions: Drug: Calcipotriol Betamethasone ointment and Calcipotriol ointment
- Calcipotriol/Betamethasone and urea cream (Sham Comparator): alcipotriol/Betamethasone ointment 1/d for 4 weeks , urea cream 1/d for 6 weeks on-demand treatment period
  Interventions: Drug: Calcipotriol Betamethasone ointment and Urea Cream
- Calcipotriol/Betamethasone (Active Comparator): Calcipotriol/Betamethasone ointment 1/d for 4 weeks, Calcipotriol/Betamethasone ointment 1/d for 6 weeks on-demand treatment period
  Interventions: Drug: Calcipotriol Betamethasone ointment

INTERVENTIONS:
Drug: Calcipotriol Betamethasone ointment and Calcipotriol ointment
  Arms: Calcipotriol/Betamethasone and Calcipotriol
Drug: Calcipotriol Betamethasone ointment
  Arms: Calcipotriol/Betamethasone
Drug: Calcipotriol Betamethasone ointment and Urea Cream
  Arms: Calcipotriol/Betamethasone and urea cream

SUMMARY:
Evaluate the efficacy and safety of Calcipotriol Betamethasone Ointment and Calcipotriol Ointment in sequential therapy

DETAILED DESCRIPTION:
1.240 subjects will be randomized 1:1:1 divided into the 3 groups 2.Week0 to Week4,each group were treated with Calcipotriol Betamethasone Ointment 3.Week4 to Week12, the there group were respectively treated with Calcipotriol Betamethasone Ointment,Calcipotriol Ointment and Urea Cream 4.The efficacy and safety were evaluated at the baseline, as well as 1, 4, 8 and 12 weeks after the beginning of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who signed Informed Consent Form；
2. Male or female subjects 18-65 years of age；
3. Clinically confirmed diagnosis of plaque psoriasis as per the diagnostic criteria for psoriasis vulgaris specified in Clinical Dermatology.
4. Involved area 1-10% of the body surface area.

Exclusion Criteria:

1. Incompliance with the diagnosis of plaque psoriasis or plaque area > 10% of the body surface area.
2. Erythrodermic psoriasis, psoriasis arfhropathica or pustular psoriasis;
3. Known allergy to any component of the test or control drug；
4. Concomitant allergic skin disease such as eczema， contact dermatitis and urticaria, or other serious and/or extensive skin disease；
5. Systemic medication or ultraviolet therapy for psoriasis within 4 weeks prior to study initiation；
6. Topical use of external drug for psoriasis within 2 weeks prior to study initiation；
7. Women of child-bearing potential who are pregnant, plan to become pregnant during study or are lactating；
8. Glucocorticoid or immunodepressant, or hypoleukemia due to tumor or chemotherapy within the last 4 weeks；
9. Serious life-threatening condition that allows a life expectancy of less than 2 months；
10. Inability to guarantee taking medications and completing visits as scheduled during the study;
11. Serious infection that is not suitable for external treatment；
12. Any other condition that the investigator deems unsuitable for entering the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index 50 ,75 and 90 | week0 and week12

SECONDARY OUTCOMES:
Time to recurrence | Any Point In Time after 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China